CLINICAL TRIAL: NCT06053476
Title: Optimal Postoperative Chest Tube and Pain Management in Patients Surgically Treated for Primary Spontaneous Pneumothorax (Pneumotrial); a Randomized Controlled Trial
Brief Title: Optimal Postoperative Chest Tube and Pain Management in Patients Surgically Treated for Primary Spontaneous Pneumothorax (Pneumotrial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maxima Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Quirine van Steenwijk, Coordinating Investigator, MD, Maxima Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NL84451.015.23
Record Dates: First submitted 2023-09-12; First posted 2023-09-25 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Pneumothorax, Primary Spontaneous; VATS; Pain, Postoperative; Locoregional Anaesthesia; Thoracic Epidural; Chest Tube Drainage
MeSH Terms: conditions — Pneumothorax; Pain, Postoperative | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Chest tube duration at least 3 days plus TEA (Active Comparator)
  Interventions: Procedure: Thoracic epidural analgesia; Procedure: Late chest tube removal
- Chest tube duration at least 3 days plus single-shot PVB (Experimental)
  Interventions: Procedure: Single-shot paravertebral block; Procedure: Late chest tube removal
- Early chest tube removal plus TEA (Experimental)
  Interventions: Procedure: Thoracic epidural analgesia; Procedure: Early chest tube removal
- Early chest tube removal plus single-shot PVB (Experimental)
  Interventions: Procedure: Single-shot paravertebral block; Procedure: Early chest tube removal

INTERVENTIONS:
Procedure: Thoracic epidural analgesia — After correct placement of the epidural catheter, a local anaesthetic (ropivacaine, levobupivacaine or bupivacaine) will be started and, according to in house protocols, an opioid will be added to the epidural solution. A provisional stop of the administration of the epidural infusion is planned after 48 hours (on the second postoperative day).
  Arms: Chest tube duration at least 3 days plus TEA; Early chest tube removal plus TEA
Procedure: Single-shot paravertebral block — At the beginning of surgery, before pleurectomy, a single shot PVB will be placed at 10 levels (T2-T11) by the surgeon with Ropivacaine 7.5mg/mL and 2-3mL per site under direct thoracoscopic vision. The injection site will be chosen at the paravertebral space, just lateral adjacent to the sympathetic trunk.
  Arms: Chest tube duration at least 3 days plus single-shot PVB; Early chest tube removal plus single-shot PVB
Procedure: Late chest tube removal — Postoperatively, the chest tube is connected to a Thopaz+ system (Medela inc.) and installed to -2 or -5 cm H2O.
  The chest tube will be left in place during a fixed period of 3 postoperative days. The chest tube will be removed at the earliest at POD 3 in case the following criteria are met:
  1. The patient is lucid and capable of sitting up straight in bed on his/her own
  2. No air leakage indicated by the Thopaz+ system during at least 4 hours, or <15 mL/min air leakage during at least 6 hours
  3. Postoperative X ray (performed at least 4 hours after surgery or ultimately performed the morning of POD1) demonstrating complete lung expansion at the level of the hilum.
  4. Absence of bloody drainage by the Thopaz+ system
  Arms: Chest tube duration at least 3 days plus TEA; Chest tube duration at least 3 days plus single-shot PVB
Procedure: Early chest tube removal — Postoperatively, the chest tube is connected to a Thopaz+ system (Medela inc.) and installed to -2 or -5 cm H2O.
  The chest tube will be removed at the earliest at 4 hours postoperatively in case the following criteria are met:
  1. The patient is lucid and capable of sitting up straight in bed on his/her own
  2. No air leakage indicated by the Thopaz+ system during at least 4 hours, or <15 mL/min air leakage during at least 6 hours
  3. Postoperative X ray (performed at least 4 hours after surgery or ultimately performed the morning of POD1) demonstrating complete lung expansion at the level of the hilum.
  4. Absence of pure blood drainage by the Thopaz+ system
  Arms: Early chest tube removal plus TEA; Early chest tube removal plus single-shot PVB

SUMMARY:
Guidelines lack high quality evidence on optimal postoperative chest tube and pain management after surgery for primary spontaneous pneumothorax (PSP). This results in great variability in postoperative care and length of hospital stay (LOS). Chest tube and pain management are prominent factors regarding enhanced recovery after thoracic surgery, and in standardised care they are crucial to improve quality of recovery and decrease LOS.

Historically, postoperative chest tubes are left in place for at least a fixed number of 3-5 days, irrespective of absence of air leakage. This period was deemed necessary for adequate pleurodesis and prevention of recurrence. However, it is suggested that removal on the same day of surgery is safe and associated with a reduced LOS.

Regarding postoperative pain management, thoracic epidural analgesia (TEA) is the gold standard for postoperative pain management following video-assisted thoracic surgery (VATS). Although the analgesic effect of TEA is clear, it is associated with hypotension and urinary retention. Therefore, unilateral regional techniques, such as paravertebral blockade (PVB), are developed.

The investigators hypothesize that early chest tube removal accompanied by a single-shot paravertebral blockade (PVB) for analgesia is safe regarding pneumothorax recurrence and non-inferior regarding pain, but superior regarding LOS when compared to standard conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients operated for PSP
* Age ≥ 16 years
* Able to read and understand the Dutch language
* Mentally able to provide informed consent
* Patients should have a preoperative chest CT scan in order to exclude evident secondary pneumothorax. Previously made CT scans, within a time range of maximum 5 years, are accepted. The identification of blebs or bullae on CT scan is not defined as secondary pneumothorax.

Exclusion Criteria:

* Previous ipsilateral thoracic surgery (except diagnostic thoracoscopy only) or ipsilateral thoracic radiotherapy
* Underlying lung disease that provoked the pneumothorax (secondary pneumothorax): genetically proven Birt-Hogg-Dubé syndrome, periodic pneumothorax in female patients in reproductive age with known endometriosis (or known catamenial pneumothorax), pulmonary cystic fibrosis, active pneumonia, lung fibrosis, chronic obstructive pulmonary disease (COPD), pulmonary ipsilateral malignancy
* Contra-indications for TEA (infection at skin site, increased intracranial pressure, non-correctable coagulopathy, sepsis and mechanical spine obstruction)
* Patients chronically (>3 months) using opioids will be excluded since postoperative baseline opioid requirement will be higher and TEA remains the preferred technique for these patients
* Allergic reactions to analgesics used in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | Until 1 year follow-up
  Safety outcome: absolute number of patients with recurrence (maximum allowable difference between early and late chest tube removal groups of 9 recurrences) defined as having an ipsilateral recurrent pneumothorax after chest tube removal, confirmed by X-ray or CT within 1-year, requiring reintervention (either tube thoracostomy or reoperation) or hospital readmission.
Pain score | Postoperative day 0-3
  Proportion of pain scores ≥4 as assessed by the numerical rating scale (NRS), defined as the number of NRS scores ≥4 divided by the total number of NRS measurements. NRS score is measured from 0 until 10; lowest value signifying no pain and highest value signifying worst pain.
Postoperative length of stay (LOS) | 30 postoperative days
  the total number of in-hospital days including readmissions due to complications or recurrence within 30 postoperative days (POD). The day of surgery will be POD 0.

SECONDARY OUTCOMES:
Quality of Recovery (QoR) | until 4 weeks follow-up
  QoR measured with the QoR-15 questionnaire on postoperative 1 and 2 (maximum score of 150, the higher the score the better the outcome)
Quality of Life (QoL) | until 1 year follow-up
  QoL will be measured using the EORTC Core Quality of Life questionnaire (EORTC QLQ-C30). This 33-item questionnaire incorporates functional scales, symptom scales and overall health status. The scale range from 0 to 100; a higher score represents a higher response level.
Postoperative complications | until 4 weeks follow-up
  according to the Clavien-Dindo classification
Postoperative chest tube drainage during hospitalisation | 30 postoperative days
  Total number of postoperative days with a chest tube. The day of surgery is day 0.
Cumulative use of opioids and analgesics | postoperative day 0-4 and the use at 4 weeks follow-up
  total opioid and non-opioid consumption as supplementary analgesic requirement
degree of mobility | postoperative day 0-4
  4-point scale: on the bed (1), to the chair (2), to the toilet (3), outside the patient's hospital room(4)
Health status | until 1 year follow-up
  Health status will we measured using the EuroQol-5D (EQ-5D) tool. This tool incorporates 5 aspects regarding health. The scale range from 0 to 100; a higher score represents a higher health status.
patient satisfaction | postoperative day 0-4
  5-point Likert scale: not at all satisfied, slightly satisfied, neutral, very satisfied and extremely satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Maxima MC, Veldhoven, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data will become available for non-commercial scientific research (open access) after a period of 12 months after the last data collection. Data request can be done by contacting the PI.
Supporting Information: Study Protocol, SAP, ICF